CLINICAL TRIAL: NCT02104674
Title: A PHASE III, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED STUDY TO EVALUATE THE EFFICACY AND SAFETY OF LEBRIKIZUMAB IN ADULT PATIENTS WITH MILD TO MODERATE ASTHMA
Brief Title: A Study Evaluating the Efficacy and Safety of Lebrikizumab in Adult Patients With Mild to Moderate Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WA29249
Record Dates: First submitted 2014-03-26; First posted 2014-04-04 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — lebrikizumab; montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Other: placebo
- Singulair (montelukast) (Active Comparator)
  Interventions: Drug: montelukast [Singulair]
- lebrikizumab (Experimental)
  Interventions: Drug: lebrikizumab

INTERVENTIONS:
Drug: lebrikizumab — Given SC on Days 1, 29, and 57
  Arms: lebrikizumab
Drug: montelukast [Singulair] — 10 mg given orally once daily for 12 weeks
  Arms: Singulair (montelukast)
Other: placebo — SC injection given on Days 1, 29, and 57
  Arms: Placebo

SUMMARY:
This Phase III, randomized, double-blind, placebo-controlled, multicenter study will assess the efficacy and safety of lebrikizumab in adult patients with mild to moderate asthma treated with short-acting beta-agonist (SABA) therapy alone. Patients will be randomized in a 1:1:1 ratio to receive either blinded lebrikizumab or placebo treatment by subcutaneous (SC) injection (every 4 weeks for a total of 3 doses) or open-label treatment with Singulair (Montelukast; 10 mg daily). Time on study treatment will last 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years old at study start
* Asthma diagnosis for >/= 12 months prior to study start
* Bronchodilator response at screening
* Pre-bronchodilator FEV1 of 60% - 85% predicted at both screening visits 2 and 3
* No other clinically significant lung disease as confirmed by chest X-ray or computed tomography (CT) scan
* Stable and symptomatic asthma during the screening period
* Use of effective contraception, as defined by the protocol, until 24 weeks after the last dose

Exclusion Criteria:

* Maintenance of corticosteroid therapy, defined as daily or alternate-day oral corticosteroid maintenance therapy within 3 months prior to study start
* Treatment with systemic or inhaled corticosteroids within 4 weeks prior to study start or during the screening period for any reason, including an acute exacerbation event
* Treatment with a leukotriene receptor antagonist (LTRA), long-acting beta-agonist (LABA) long-acting muscarinic antagonist (LAMA), zileuton, roflumilast, or theophylline within 2 weeks prior to study start
* Documented prior treatment failure with Montelukast
* Treatment with intra-articular corticosteroids within 4 weeks prior to study start or during the screening period or anticipated need for intra articular corticosteroids during the course of the study
* Any infection requiring hospital, IV or IM antibiotic treatment or any respiratory infection within 4 weeks of study start. Any infection requiring oral antibiotic treatment within 2 weeks of study start, or any parasitic infection within 6 months of study start
* Clinically significant abnormality found during screening or clinically significant medical disease that is uncontrolled despite treatment that is likely, in the opinion of the investigator, to impact the patient's ability to participate in the study, or impact the study assessments
* History of interstitial lung disease, chronic obstructive pulmonary disease (COPD), or other clinically significant lung disease other than asthma
* History of alcohol or drug abuse that would impair or risk the patient's full participation in the study, in the opinion of the investigator
* Current or history of smoking (> 10 pack-years), or unwillingness to abstain from smoking for the duration of the study
* Past and/or current use of any anti-IL-13 or anti- IL4/IL-13 therapy, including lebrikizumab
* Use of a licensed or investigational monoclonal antibody other than anti IL-13 or anti-IL-4/IL-13, including, but not limited to, omalizumab, anti-IL-5, or anti IL-17, within 6 months or 5 drug half-lives prior to Visit 1 (whichever is longer) or during screening
* Use of a systemic immunomodulatory or immunosuppressive therapy within 3 months or 5 drug half-lives prior to study start or during screening
* Use of other investigational therapy within 4 weeks or 5 drug half-lives prior to study start (whichever is longer) or during screening
* Initiation of or change in allergen immunotherapy within 3 months prior to study start or during screening
* Receipt of a live attenuated vaccine within 4 weeks prior to study start of during screening
* Pregnancy or breast feeding
* Body mass index > 38 kg/m2
* Body weight < 40 kg
* History of bronchial thermoplasty

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2014-06; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Absolute change in pre-bronchodilator forced expiratory volume in 1 second (FEV1) | From Baseline to Week 12

SECONDARY OUTCOMES:
Relative change in morning pre-bronchodilator peak expiratory flow (PEF) | From Baseline to Week 12
Time to treatment failure | From Baseline to Week 12
Change in asthma rescue medication use | From Baseline to Week 12
Incidence of adverse events | Approximately 20 weeks
Pharmacodynamics: Relative change in fractional exhaled nitric oxide (FeNO) | From Baseline to Week 12
Pharmacodynamics: Change in blood eosinophil count | From Baseline to Week 12
Pharmacokinetics: Maximum serum lebrikizumab concentration after the first dose (Cmax) | Week 1
Change in patient-reported outcome, as measured by the Standardized Asthma Quality of Life Questionnaire (AQLQ(S)) | From Baseline to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (95):
- United States (49):
  - Birmingham, Alabama
  - Flagstaff, Arizona
  - Scottsdale, Arizona
  - Alhambra, California
  - Anaheim, California
  - Los Angeles, California
  - Napa, California
  - Rancho Mirage, California
  - Redwood City, California
  - Stockton, California
  - Upland, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Waterbury, Connecticut
  - Cooper City, Florida
  - Kissimmee, Florida
  - New Port Richey, Florida
  - Winter Park, Florida
  - Columbus, Georgia
  - Duluth, Georgia
  - Normal, Illinois
  - Oak Lawn, Illinois
  - River Forest, Illinois
  - Avon, Indiana
  - Louisville, Kentucky
  - Minneapolis, Minnesota
  - Plymouth, Minnesota
  - St Louis, Missouri
  - Papillion, Nebraska
  - Ocean City, New Jersey
  - Rochester, New York
  - The Bronx, New York
  - Hendersonville, North Carolina
  - High Point, North Carolina
  - Oklahoma City, Oklahoma
  - Medford, Oregon
  - Portland, Oregon
  - Greer, South Carolina
  - Boerne, Texas
  - Dallas, Texas
  - Houston, Texas
  - Humble, Texas
  - McKinney, Texas
  - San Antonio, Texas
  - Tomball, Texas
  - Waco, Texas
  - Fairfax, Virginia
  - Henrico, Virginia
  - Greenfield, Wisconsin
- Brazil (4):
  - Rio de Janeiro, Rio de Janeiro
  - Porto Alegre, Rio Grande do Sul
  - Florianópolis, Santa Catarina
  - Santo André, São Paulo
- Bulgaria (6):
  - Gabrovo
  - Razgrad
  - Rousse
  - Sofia
  - Varna
  - Veliko Tarnovo
- Canada (2):
  - Brampton, Ontario
  - Toronto, Ontario
- Czechia (4):
  - Jablonec nad Nisou
  - Jindřichův Hradec
  - Karlovy Vary - Stará Role
  - Strakonice
- Tbilisi, Georgia
- New Zealand (2):
  - Auckland
  - Beckenham
- Poland (7):
  - Bialystok
  - Krakow
  - Lodz
  - Lublin
  - Poznan
  - Tarnów
  - Wroclaw
- Puerto Rico (2):
  - Caguas
  - San Juan
- Romania (5):
  - Bucharest
  - Cluj-Napoca
  - Iași
  - Oradea
  - Timișoara
- Russia (5):
  - Moscow
  - Ryazan
  - Saint Petersburg
  - Saratov
  - Yekaterinburg
- Spišská Nová Ves, Slovakia
- South Africa (6):
  - Cape Town
  - Johannesburg
  - Lyttleton
  - Parow
  - Pretoria Gauteng Province
  - Soweto
- Manchester, United Kingdom

REFERENCES:
- [Derived] Korenblat P, Kerwin E, Leshchenko I, Yen K, Holweg CTJ, Anzures-Cabrera J, Martin C, Putnam WS, Governale L, Olsson J, Matthews JG. Efficacy and safety of lebrikizumab in adult patients with mild-to-moderate asthma not receiving inhaled corticosteroids. Respir Med. 2018 Jan;134:143-149. doi: 10.1016/j.rmed.2017.12.006. Epub 2017 Dec 13. PMID 29413502